CLINICAL TRIAL: NCT01378585
Title: A Randomized, Double Blind, Placebo Controlled, Cross-over, and Fixed Dose Study to Evaluate the Safety and Efficacy of DLBS1033 in Healthy Subjects
Brief Title: Safety and Efficacy of DLBS1033 in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS1033
Record Dates: First submitted 2011-06-06; First posted 2011-06-22 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: DLBS1033; safety; fibrinolytic; fibrinogenolytic; antiplatelet
MeSH Terms: interventions — DLBS 1033

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Treatment 1 (Experimental): Test drug treatment: 3 x 490 mg DLBS1033 daily
  Interventions: Drug: DLBS1033
- Treatment 2 (Placebo Comparator): Placebo treatment: 3 x 1 tablet daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DLBS1033 — 3 x 490 mg DLBS1033 daily
  Arms: Treatment 1
Drug: Placebo — 3 x 1 tablet daily
  Arms: Treatment 2

SUMMARY:
The objective of this study are:

1. To evaluate the safety of DLBS1033 in comparison with placebo in healthy adult subject
2. To evaluate the efficacy of DLBS1033 in comparison with placebo in healthy adult subject

DETAILED DESCRIPTION:
This study is a 2-arm, randomized, double-blind, placebo controlled, cross-over study with a fixed dose regimen. The study will involve twenty (20) healthy subjects. The study will be a comparative study of safety and efficacy of DLBS1033 with placebo. Each study period will consist of 14 days treatment with a 2-week wash-out period in between. The evaluation of safety parameters will be performed at Day 1 (baseline), 7, and 14; while the efficacy parameters will be performed at Day 1, 2, 7, and 14.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 50 year-old at screening
* Having good and stable health judged on the basis of medical history, physical examination, and routine laboratory
* Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study

Exclusion Criteria:

* Participating in other clinical trial within 4 weeks prior to screening
* Had a major surgical procedure or dental procedure within 4 weeks prior to screening
* History of any of the following medical conditions: haemophilia, past medical history of haemorrhagic stroke, acid peptic disease, easy bruising and frequent external bleeding
* Any other known current medical condition, which is judged by the investigator could jeopardize subject's health or interfere with the study evaluation
* Being on regular medication(s), including traditional medicine(s)
* Pregnant or lactating women (urinary pregnancy test will be applied to women subjects during screening and just before treatment in each periods)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety | 14 days
  routine hematology (Hb, Ht, RBC, WBC, Platelet), erythrocyte sedimentation rate (ESR), liver function (ALT, AST, Gamma-GT, alkaline phosphatase), renal function (ureum, creatinine), lipid profile (total cholesterol, triglyceride, LDL-C, HDL-C), fasting blood glucose, routine urine parameters (glucose, bilirubin, ketones, specific gravity, blood, urinary pH, proteins, urobilinogen, nitrites, leucocyte esterase, and urine sediment), stool occult blood, ECG examination, clinical / physical examination

SECONDARY OUTCOMES:
Fibrinogen level | Day 1, 2, 7, and 14 of treatment
Thrombin time (TT) | Day 1, 2, 7, and 14 of treatment
prothrombin time (PT) | Day 1, 2, 7, and 14 of treatment
activated-partial thromboplastin time (aPTT) | Day 1, 2, 7, and 14 of treatment
Number of subjects with adverse events | Day 1 and 7 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Danang A Yunaidi, Dr, Principal Investigator — PT Equilab International
Locations (1):
- PT Equilab International, Jakarta, Jakarta Special Capital Region, Indonesia